CLINICAL TRIAL: NCT05545462
Title: Comparison Of Doxycycline And Common Salt (TableCooking) For Treatment Of Umbilical Granuloma In Children: A Randomised Control Trial
Brief Title: Comparison Of Doxycycline And Common Salt For Treatment Of Umbilical Granuloma: A Randomised Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr.M. Awais, Dr. Muhammad Awais, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 356/SZABMU/MS-2017
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Umbilical Granuloma
MeSH Terms: interventions — Doxycycline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COMPARISON OF DOXYCYCLINE AND COMMON SALT FOR TREATMENT OF UMBILICAL GRANULOMA IN CHILDREN (Experimental): to study the comparison of doxycycline and common salt for the treatment of umbilical granuloma to check which is more effective safe timesaving and can be performed by even parents it showed that common salt is more effective than doxycycline
  Interventions: Drug: Doxycyclin
- COMPARISON BETWEEN COMMON SALT AND SOXYCYLIN FOR TREATMENT OF UMBILICAL GRANULOMA (Experimental): to study the comparison of doxycycline and common salt for the treatment of umbilical granuloma to check which is more effective safe timesaving and can be performed by even parents it showed that common salt is more effective than doxycycline
  Interventions: Other: COMMON SALT

INTERVENTIONS:
Drug: Doxycyclin — THE USE OF DOXYCYCLIN POWDER IN THE TREATMENT OF UMBILICAL GRANULOMA
  Other Names: COMMON SALT
  Arms: COMPARISON OF DOXYCYCLINE AND COMMON SALT FOR TREATMENT OF UMBILICAL GRANULOMA IN CHILDREN
Other: COMMON SALT — THE USE OF COMMON SALT IN TREATMENT OF UMBILICAL GRANULOMA
  Arms: COMPARISON BETWEEN COMMON SALT AND SOXYCYLIN FOR TREATMENT OF UMBILICAL GRANULOMA

SUMMARY:
it is the study for the disease called umbilical granuloma to look for the better treatment option which can be performed by healthcare physicians and local nurses and even parents

DETAILED DESCRIPTION:
umbilical granuloma is a condition for which multiple treatments are available those including interventional and non interventional, most of the treatments are performed by the health care physician like application of silver nitrate cryotherapy, electrocautery, double ligation.

the main goal of this study is to prefer those method or drugs which could be safely used by the nurses the health care personal and even by parents at home with fewer side effects

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Neonates and infants (age<1yr)
  2. Both genders
  3. Confirmed by ultrasonography and sinography (if applicable)

Exclusion Criteria:

* 1. If any treatment is already given 2. Patient lost in follow up 3. Refusal

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison Of Doxycycline And Common Salt (TableCooking) For Treatment Of Umbilical Granuloma In Children: A Randomised Control Trial | 1 year
  for the treatment of Umbilical Granuloma multiple treatment options are available. and we have studied about the two methods the common salt any doxycycline The use of common salt to treat umbilical granuloma is a simple, highly effective, and inexpensive with minimum complications or relapse as compared to doxycycline. Treatment can be performed by physicians, nurses, primary health-care staff in remote areas, and even by parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan institute of medical Sciences/ Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan